CLINICAL TRIAL: NCT02895165
Title: An Italian Multicenter Prospective Cohort Study on Fertility Preservation and Pregnancy Issues in Young Breast Cancer Patients: PREgnancy and FERtilty (PREFER)
Brief Title: PREgnancy and FERtility Registry
Acronym: PREFER
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Collaborators: Clinical Research Technology S.r.l. (Industry)
Responsible Party: Principal Investigator, Lucia Del Mastro,MD, MD, IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Other Study IDs: 001377;000650
Record Dates: First submitted 2016-08-22; First posted 2016-09-09 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Breast Neoplasms; Pregnancy; Fertility Preservation
Keywords: breast neoplasms; fertility preservation; pregnancy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The PREgnancy and FERtility (PREFER) study is a comprehensive program aiming to optimize care and improve knowledge around the topics of fertility preservation and pregnancy issues in young breast cancer patients. The program was initiated at the National Institute for Cancer Research, IRCCS AOU San Martino - IST in Genova (Liguria Region, Italy) and then it has been spread to other Italian Institutions under the umbrella of the Gruppo Italiano Mammella (GIM) study group. It is composed of two distinctive studies, one assessing fertility (i.e. PREFER-FERTILITY) and the other pregnancy (PREFER-PREGNANCY) issues. Hence, two different study protocols were developed under the umbrella of the PREFER registry.

PREFER-FERTILITY aims to obtain and centralize data about the preferences and choices of young cancer patients on the fertility preservation strategies available in Italy. Furthermore, it aims to assess the outcomes of patients undergoing one or more strategies for fertility preservation in terms of success of the techniques (i.e. recovery of ovarian function, number of cryopreserved oocytes, post-treatment pregnancies) and safety (i.e. long-term survival outcomes).

PREFER-PREGNANCY has two main objectives: 1) to obtain and centralize data on the management of breast cancer diagnosed during pregnancy, the obstetrical and paediatric care of children born after prior in utero exposure to anticancer treatments, and the long-term survival outcomes of these patients; 2) to obtain and centralize data on the clinical outcomes of breast cancer survivors that achieve a pregnancy after prior diagnosis and treatment of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer diagnosis
* age between18 and 45 years (only for PREFER-FERTILITY)
* have not received any radiation or chemotherapy for cancer before enrolment (only for PREFER-FERTILITY)
* absence of metastatic disease (only for PREFER-FERTILITY)
* diagnosis of breast cancer during pregnancy or within 1 year from the end of pregnancy or pregnancy after prior diagnosis and treatment for breast cancer (only for PREFER-PREGNANCY)
* informed consent

Exclusion Criteria:

* inability to provide written informed consent
* stage IV disease at diagnosis (only for PREFER-FERTILITY)
* serious psychiatric disorders

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young breast cancer patients facing fertility and pregnancy issues
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-11; Primary Completion 2027-11 (Estimated); Study Completion 2032-11 (Estimated)

PRIMARY OUTCOMES:
Rate of patients interested in the available strategies for fertility preservation | 15 years
  Assessed through medical records
Rate of patients undergoing the different strategies for fertility preservation | 15 years
  Assessed through medical records
Type of strategies for fertility preservation proposed by oncologists | 15 years
  Assessed through medical records
Reasons for refusal of the available strategies for fertility preservation | 15 years
  Assessed through an open questionnaire
Type of anticancer therapies administered during pregnancy | 15 years
  Assessed through medical records
Safety: pregnancy complications | 15 years
  Assessed through medical records
Safety: incidence of adverse events | 15 years
  Assessed through medical records
Disease-free survival | 15 years
Overall survival | 15 years

SECONDARY OUTCOMES:
Success of the available strategies for fertility preservation: rate of recovery of ovarian function after antitumor treatments | 15 years
Success of the available strategies for fertility preservation: number of oocytes collected and cryopreserved | 15 years
Success of the available strategies for fertility preservation: number of pregnancies achieved after breast cancer treatments | 15 years
Serum hormonal changes during chemotherapy and study follow up | 15 years
  FSH (follicle stimulating hormone), estradiol and AMH (anti-mullerian hormone) serum levels assessed at baseline, during chemotherapy, at the end of chemotherapy and every six months thereafter
Obstetrical and paediatric care of children born after prior in utero exposure to anticancer treatments | 15 years
  Assessed using obstetric and paediatric medical records
Obstetrical and paediatric care of children born in breast cancer survivors | 15 years
  Assessed using obstetric and paediatric medical records

CONTACTS AND LOCATIONS:
Locations (23):
- Italy (23):
  - Presidio Ospedaliero 'Antonio Perrino', Brindisi, BR
  - AOU di Cagliari Strada, Monserrato, Cagliari
  - Azienda Ospedaliera S. Croce e Carle, Cuneo, CN
  - Arcispedale S. Anna - A.O.U. di Ferrara, Cona, FE
  - Irccs Aou San Martino - Ist, Genoa, GE
  - Ospedale Vito Fazzi, Lecce, LE
  - Ospedale Unico Versilia, Lido di Camaiore, LU
  - Azienda Ospedaliera Carlo Poma, Mantova, MN
  - Ospedale 'Guglielmo da Saliceto', Piacenza, PC
  - Fondazione S. Maugeri IRCCS, Pavia, PV
  - Azienda Ospedaliera S. Carlo, Potenza, PZ
  - Istituto Regina Elena per lo studio e la cura dei tumori, Roma, RM
  - Azienda Ospedaliera n. 1 - Annunziata, Sassari, SS
  - Fondazione del Piemonte per l'Oncologia - IRCC di Candiolo, Candiolo, TO
  - AOU SM Misericordia, Udine, UD
  - Ospedale Sacro Cuore Don Calabria, Negrar, VE
  - Ospedale Cardinal Massaia, Asti
  - A.O.U. Federico II, Napoli
  - Istituto Nazionale dei Tumori - Fondazione G.Pascale, Napoli
  - Ospedale Santa Maria della Misericordia, Perugia
  - AOU Pisana - Ospedale S. Chiara, Pisa
  - Arcispedale Santa Maria Nuova di Reggio Emilia, Reggio Emilia
  - ASS1 Triestina, Trieste

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lambertini M, Anserini P, Fontana V, Poggio F, Iacono G, Abate A, Levaggi A, Miglietta L, Bighin C, Giraudi S, D'Alonzo A, Blondeaux E, Buffi D, Campone F, Merlo DF, Del Mastro L. The PREgnancy and FERtility (PREFER) study: an Italian multicenter prospective cohort study on fertility preservation and pregnancy issues in young breast cancer patients. BMC Cancer. 2017 May 19;17(1):346. doi: 10.1186/s12885-017-3348-8. PMID 28526012